CLINICAL TRIAL: NCT05485064
Title: Moderate Sedation Combined With Acupuncture Anesthesia in Gastroscopy and Colonoscopy on Screening Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jixiangyu, associate chief physician, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QYFYKYLL 916711920
Record Dates: First submitted 2022-07-29; First posted 2022-08-03 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Gastrointestinal Endoscopy
Keywords: eletroacupuncture; moderate sedation; remimazolam; transcutaneous electrical acupuncture point stimulation
MeSH Terms: interventions — Fentanyl; remimazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: During the examination, the acupuncture position was blocked to ensure that the acupuncture position was not visible; except for researcher 1, the only researcher who knew about the grouping of patients,All trial-related data were recorded by researcher 2 , and researcher 1 was responsible for patients'sedation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electroacupuncture(transcutaneous electrical acupuncture point stimulation )and remimazolam (Experimental): The investigator 1 combine electroacupuncture(transcutaneous acupoint electrical stimulation ) with remimazolam to sedate patients moderately to finish gastroscopy and colonoscopy.
  Interventions: Procedure: eletroacupuncture(transcutaneous electrical acupuncture point stimulation ); Drug: remimazolam
- placebo needle and remimazolam (Experimental): The investigator 1 combine placebo needle with remimazolam to sedate patients moderately to finish gastroscopy and colonoscopy.
  Interventions: Drug: placebo needle; Drug: remimazolam
- fentanyl and remimazolam (Experimental): The investigator 1 combine fentanyl with remimazolam to sedate patients moderately to finish gastroscopy and colonoscopy.
  Interventions: Drug: fentanyl; Drug: remimazolam

INTERVENTIONS:
Drug: fentanyl — The investigator 1 use fentanyl to sedate patients coordinate with remimazolam
  Arms: fentanyl and remimazolam
Procedure: eletroacupuncture(transcutaneous electrical acupuncture point stimulation ) — The investigator 1 use electroacupunture(transcutaneous electrical acupuncture point stimulation )to coordinate with remimazolam
  Arms: electroacupuncture(transcutaneous electrical acupuncture point stimulation )and remimazolam
Drug: placebo needle — The investigator 1 use placebo needle to sedate patients coordinate with remimazolam
  Arms: placebo needle and remimazolam
Drug: remimazolam — The investigator 1 use remimazolam to sedate patients coordinate with eletroacupuncture(transcutaneous electrical acupuncture point stimulation )or placebo needle

SUMMARY:
The purpose of this study is mainly about the feasibility and rationality of moderate sedation combined with acupuncture anesthesia in the application of gastroscopy and colonoscopy ,Then we evaluate the effectiveness and advantages of the combination of acupuncture anesthesia and drug anesthesia.

DETAILED DESCRIPTION:
With the increase of the proportion of the patients who crave for performing painless gastroscopy and colonoscopy in recent years, it is crucial to seek a more secure and effective method of anesthesia or sedation. At present, the universal anesthetic method on gastroscopy and colonoscopy in China is the general anesthesia without intubation which usually uses propofol and opioid analgesics,Although the satisfaction of patients is high, the incidence of anesthesia-related complications and drug-related adverse reactions is high .The incidence of adverse events during the gastroscopy and colonoscopy is high, and the medical expense of anesthesia is high. At present, more than 2/3 of the patients undergo painless gastroscopy or colonoscopy are middle-aged and elderly patients, so the overdose which prolongs the recovery time、discharge time of patients and reduces the recovery quality of patients is common. The moderate sedation, which fundmentally does not affect hemodynamics、autonomous respiration and protective reflexes, is incomparable to general anesthesia . And acupuncture anesthesia also acts as a safe anesthetic method can provide safer analgesic effect.Theoretically，the combination of both of them is a relatively perfect and safe painless method.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. Patients with ASA grade I-III
3. A sufficient level of education to understand study procedures and can communicate with investigators.

Exclusion Criteria:

1. Patients with serious systemic diseases such as severe cardiopulmonary disease or hepatic diseases or renal diseases.
2. Patients under the age of 18.
3. Patients who did not sign the informed consent form.
4. Patients who have a history of alcohol abuse or drug abuse.
5. People who are allergic to anesthetic related ingredients, such as soybeans, eggs and so on.
6. Patients with extreme fear or anxiety about acupuncture.
7. Patients with relative contraindications of gastrointestinal endoscopy.

   -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
patient satisfaction with sedation instrument，PSSI | During gastroscopy and colonoscopy
  The investigator 2 needs to use VAS scores to evaluate satisfaction about sedation feeling when they accepted gastroscopy and colonoscopy .The score ranges from 0 to10 and need patients evaluate it by themself when the gastroscopy or colonoscopy were finished.The score from 0 （extremely dissatisfied）to 10（extremely satisfied）.
clinical satisfaction with sedation instrument，CSSI | During gastroscopy and colonoscopy
  The investigator 2 needs to use VAS scores to evaluate satisfaction about doctors when they carry out the operation.The score from 0 （extremely dissatisfied）to 10（extremely satisfied）.
patient's pain score | During gastroscopy and colonoscopy
  The investigator 2 needs to use VAS scores to evaluate patients' pain score .The score from 0 （extremely dissatisfied）to 10（extremely satisfied）.

SECONDARY OUTCOMES:
the extent of cardia exposure | During gastroscopy and colonoscopy
  The investigator 2 needs to record the extent of cardia exposure to evaluate these interventions'effect on gastroscopy ，the investigator 2 use the table of the extent of preventriculus exposure（score from 1 to 4，1=the extent of exposure lower than 25%；2=the extent of exposure between 25% and 50%；3=the extent of exposure between 50%and 75%；4=the extent of exposure between 75%and 100%）
adverse reactions | During gastroscopy and colonoscopy
  The investigator 2 needs to record the adverse reactions such as nausea、emesis, salivation, restlessness, and breath holding to analyze efficacy of relate treatment.
patient's recovery time | The end of gastroscopy and colonoscopy
  The investigator 2 needs to record to evaluate patient's recovery quality about patients
patient's departure time | The end of gastroscopy and colonoscopy
  The investigator 2 needs to record patient's departure time to evaluate recovery quality about patients
time to resume normal operation | The end of gastroscopy and colonoscopy
  The investigator 2 needs to record the time to resume normal operation about patient
operation time about gastrointestinal endoscopy | During gastroscopy and colonoscopy
  The investigator 2 needs to record operation time about gastrointestinal endoscopy.
heart rate | before gastrointestinal endoscopy、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy
  The investigator 2 needs to record heart rate（for example 60 times/min）before gastrointestinal endoscopy 、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy respectively.（tachycardia：heart rate is more than 100 times/min；bradycardia：heart rate is less than 60 times/min）
pulse oximetry | before gastrointestinal endoscopy、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy
  The investigator 2 needs to record pulse oximetry (for example 97% )before gastrointestinal endoscopy 、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy respectively.（hypoxemia：pulse oximetry is lower than 90%）
systolic pressure 、diastolic pressure | before gastrointestinal endoscopy、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy
  The investigator 2 needs to record systolic pressure 、diastolic pressure(for example 120/75mmHg ) before gastrointestinal endoscopy 、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy respectively.（hypertension：systolic pressure ≥140mmHg or diastolic pressure ≥90mmHg；hypotension：systolic pressure ≤90mmHg or diastolic pressure ≤60mmHg）
respiratory rate | before gastrointestinal endoscopy、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy
  The investigator 2 needs to record respiratory rate(for example 15 times/min)before gastrointestinal endoscopy 、during gastrointestinal endoscopy and the end of gastrointestinal endoscopy respectively.（tachypnea：respiratory rate is more than 20 times/min；bradypnea：respiratory rate is less than 12 times/min）

CONTACTS AND LOCATIONS:
Locations (1):
- Jixiangyu, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF

REFERENCES:
- [Background] Eberl S, Monteiro de Olivera N, Bourne D, Streitberger K, Fockens P, Hollmann MW, Preckel B. Effect of electroacupuncture on sedation requirements during colonoscopy: a prospective placebo-controlled randomised trial. Acupunct Med. 2020 Jun;38(3):131-139. doi: 10.1136/acupmed-2017-011459. Epub 2020 Jan 22. PMID 31968988
- [Background] Yu B, Hazlewood PJ, Yin X, Li S, Yue H, Xu K, Xu S, Mi Y. Effect of electroacupuncture on discomfort during gastroscopy: a study protocol for a randomized controlled trial. Trials. 2022 Apr 27;23(1):364. doi: 10.1186/s13063-022-06165-4. PMID 35477483
- [Background] Cohen LB, Hightower CD, Wood DA, Miller KM, Aisenberg J. Moderate level sedation during endoscopy: a prospective study using low-dose propofol, meperidine/fentanyl, and midazolam. Gastrointest Endosc. 2004 Jun;59(7):795-803. doi: 10.1016/s0016-5107(04)00349-9. PMID 15173791
- [Background] Qin Z, Ding Y, Xu C, Kwong JSW, Ji Y, Wu A, Wu J, Liu Z. Acupuncture vs Noninsertive Sham Acupuncture in Aging Patients with Degenerative Lumbar Spinal Stenosis: A Randomized Controlled Trial. Am J Med. 2020 Apr;133(4):500-507.e20. doi: 10.1016/j.amjmed.2019.08.038. Epub 2019 Sep 13. PMID 31525334
- [Result] Chen JM, Li DD, Chen YS, Lian B, Wang XP, Guo YH, Xu XL, Huang P, Chen TF, Liu Y, Liu QQ. The effectiveness of electro-acupuncture combined with dyclonine hydrochloride in relieving the side effects of gastroscopy: a controlled trial. Ann Palliat Med. 2021 Mar;10(3):2958-2970. doi: 10.21037/apm-20-831. Epub 2021 Mar 1. PMID 33691439
- [Derived] Xu JH, Tan HL, Zhang LN, Zhou ZG, Yuan L, Kong LX, Song MQ, Qi LJ, Ji XY. Transcutaneous Electrical Acupoint Stimulation Combined with Moderate Sedation of Remimazolam Tosilate in Gastrointestinal Endoscopy: A Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Pain Ther. 2024 Aug;13(4):919-936. doi: 10.1007/s40122-024-00618-1. Epub 2024 Jun 18. PMID 38890239